CLINICAL TRIAL: NCT00154466
Title: An Association Study Between Cardiac Rehabilitation and Stem Cell Mobilization in Patients With Myocardial Infarction
Brief Title: Study on the Efficacy and Mechanism of Cardiac Rehabilitation for Stem Cell Mobilization and Heart Failure Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9261701248
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction, stem cell, cardiac rehabilitation
MeSH Terms: conditions — Myocardial Infarction | interventions — Cardiac Rehabilitation; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cardiac rehabilitation (Experimental): Those in the training group participated in a 3-month rehabilitation training program at an exercise intensity of 55% to 70% of peak oxygen uptake (VO2.
  Interventions: Behavioral: cardiac rehabilitation
- postinfarction patients (No Intervention): those in the nontraining group continued their usual lifestyle
- healthy controls (Placebo Comparator): Age-, weight-, and height-matched subjects without cardiovascular risk factors were selected as healthy controls.

INTERVENTIONS:
Behavioral: cardiac rehabilitation — Those in the training group participated in a 3-month rehabilitation training program at an exercise intensity of 55% to 70% of peak oxygen uptake (VO2); those in the nontraining group continued their usual lifestyle.
  Other Names: exercise training
  Arms: cardiac rehabilitation

SUMMARY:
One emerging concept is that some form of injury or inflammation is a prerequisite for the success of circulating-cell participation in differentiated tissue structure and function. Once reperfusion is achieved in acute myocardial infarction, an intense inflammatory cascade is unleashed.

The architecture of the left ventricle rearranges, leading to ventricular remodeling. The "homing process"involves stem cell migration to the sites of injury or ischemia, which provides an environment that is favorable to growth and function. This microenvironment is a stimulus for homing and differentiation of stem cells of the appropriate lineage. It increases vascular permeability and expression of adhesion proteins like integrin, along with homing receptors that facilitate the attachment, which is mediated by cell-to-cell contact and chemoattractant release from local tissue injury.The migratory capacity of stem cells might be dependent on natural growth factors such as vascular endothelial growth factor (VEGF) , stromal cell-derived factor-1 (SDF-1)and stem cell factor (SCF).The expression of VEGF ,SDF-1 and SCF is highly up-regulated in hypoxic tissue, supporting the hypothesis that these factors may represent homing signals crucial to the recruitment of circulating progenitor cells to assist the endogenous repair mechanisms in the infarcted tissue. This study will examine whether cardiac rehabilitation increases the concentration of stem cell factors released into the bloodstream and if these factors are correlated with the improvement of heart function.

DETAILED DESCRIPTION:
Exercise training has beneficial hemodynamic effects in patients with congestive heart failure.A similar benefit may be seen after MI, with an improvement in functional capacity averaging 20 percent. More important, however, is the possible effect on survival. In a meta-analysis of 24 trials examining the effect of cardiac rehabilitation after MI, there was a significant reduction in mortality with rehabilitation (odds ratio 0.81).

Previous studies focused on the effect of rehabilitation comes from the improvement of oxygen utilization in skeletal muscle. The effects on cardiac morphology and perfusion status were rather little to be addressed.

In this study, we will collect the questionaires, blood sampling for assay of stem cell factors, maximal O2 consumption, and cardiac MRI before and after cardiac rehabilitation.SDF-1 (stromal cell derived factor-1), SCF(stem cell factor), and VEGF (vasculoendothelial growth factor) will be measured by ELISA. Cardiac MRI will provide the information about (1) LV function, (2) scar size, and (3) perfusion status (dipyridamole stress MRI).

ELIGIBILITY:
Inclusion Criteria: myocardial infarction with CK more than 3000, status post revascularization therapy, clinical stable with regular follow-up at OPD, NYHA II-III -

Exclusion Criteria:sustained ventricular arrhythmia, hypertrophy cardiomyopathy, intolerance to exercise program

-

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-07; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bai-Chin Lee, MD, Principal Investigator — National Taiwan University Hospital; Ssu-Yuan Chen, MD, Principal Investigator — National Taiwan University Hospital; Wen-Yih Tseng, MD, PhD, Principal Investigator — National Taiwan University Hospital; Ming-Fong Chen, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Lee BC, Hsu HC, Tseng WY, Su MY, Chen SY, Wu YW, Chien KL, Chen MF. Effect of cardiac rehabilitation on angiogenic cytokines in postinfarction patients. Heart. 2009 Jun;95(12):1012-8. doi: 10.1136/hrt.2008.153510. Epub 2009 Mar 19. PMID 19304668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective randomised controlled study was approved by the ethics committee of the National Taiwan University Hospital. Between August 2004 and December 2005, 91 postinfarction patients were informed about the trial. Thirty-seven refused to participate and 15 did not meet the inclusion criteria.
Pre-assignment Details: Inclusion criteria:a successful primary stenting, a clinically stable course after MI, and no ischemia on exercise testing. Exclusion criteria: effort angina, Af, sustained ventricular arrhythmia, NYHA functional class IV, exercise-limiting diseases, severe pulmonary or renal disease, an implanted pacemaker, or claustrophobia.
Groups:
- Post-infarction Training: which underwent a 3-month cardiac rehabilitation program
- Post-infarction Nontraining: in which patients continued their usual lifestyle.
- Healthy Controls: For comparison of myocardial perfusion and angiogenic cytokines, 19 age-, weight-, and height-matched subjects without cardiovascular risk factors were selected as healthy controls.
Period: Overall Study
Arm/Group | Post-infarction Training | Post-infarction Nontraining | Healthy Controls
Started | 20 | 19 | 19 (Healthy controls underwent the test of myocardial perfusion only at baseline.)
Completed | 20 | 19 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Postinfarction Training Patients; Postinfarction Nontraining Patients; Healthy Controls: 39 postinfarction patients randomised to either a 3-month training group (n=20) or a nontraining group (n=19), and 19 normal controls.
- Total: Total of all reporting groups
Arm/Group | Postinfarction Training Patients | Postinfarction Nontraining Patients | Healthy Controls | Total
Number analyzed (Participants) | 20 | 19 | 19 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 19 | 58
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8) | 52 (9) | 50 (9) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 19 | 19 | 58
Region of Enrollment [Number; unit: participants]
  Taiwan | 20 | 19 | 19 | 58

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Blood Flow at Baseline and 3-month Follow-up
Description: First-pass, contrast-enhanced myocardial perfusion images acquired for 80 heart beats in the left ventricle. Short-axis views were obtained after intravenous administration of gadodiamide. Perfusion studies were performed at rest and during the stress induced by a 4 min infusion of dipyridamole at a concentration of 0.14 mg/kg of body weight per minute.To determine absolute MBF values at rest and stress status, we adopted a model-independent deconvolution method proposed by Jerosch-Herold et al, a method that was previously validated in experimental animal studies by comparison with blood-flow measurements with radiolabelled microspheres.
Time Frame: 3 months
Population: Eligible patients were randomly assigned to the training group, which underwent a 3-month cardiac rehabilitation program, or the nontraining group in which patients continued their usual lifestyle. Healthy controls underwent the test of myocardial perfusion only at baseline. The analysis was intention-to-treat.
Measure: Mean (Standard Deviation); unit: ml/min/g
Groups:
- Post-infarction Training; Post-infarction Nontraining: Eligible patients who provided written informed consent were randomly assigned to the training group, which underwent a 3-month cardiac rehabilitation program, or the nontraining group in which patients continued their usual lifestyle. At baseline and the 3-month follow-up, all patients underwent a functional evaluation that included clinical evaluation, exercise testing, cardiac magnetic resonance imaging (MRI), and measurements of plasma angiogenic cytokines levels. Both groups were receiving stable and optimal pharmacologic treatment supervised by their physicians.
Arm/Group | Post-infarction Training | Post-infarction Nontraining
Number analyzed (Participants) | 20 | 19
ml/min/g
  Change of stress MBF in the remote myocardium | 0.62 (0.83) | -0.27 (0.56)
  Change of stress MBF in the infarcted myocardium | 0.44 (0.71) | 0 (0.46)

2. Secondary Outcome: Angiogenic Cytokines at Baseline and 3-month Follow-up
Description: Angiogenic cytokines such as vascular endothelial growth factor (VEGF), stromal-derived factor-1 (SDF-1) and stem cell factor (SCF) are known to increase the formation of new vessels at ischaemic sites and thus enhance myocardial perfusion. To rule out any effect of short-term exercise on cytokines levels, blood samples were always taken after at least 72 h of physical inactivity and overnight fasting when the subject had rested in the sitting position for at least 10 min. The plasma samples were immediately frozen and stored at -70°C. High-sensitivity ELISA (Bender MedSystems, R&D) were used to measure plasma levels of SCF, SDF-1 and VEGF according to the manufacturer's protocols.
Time Frame: 3 months
Population: We calculated that we would need 18 patients in each group to achieve a power of at least 80% to detect a 20% difference in MBF change between study groups, with a two-sided significance level of p<0.05, and a 20% increase for the stress MBF change from baseline to 3 months' follow-up. The analysis was intention-to-treat.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Post-infarction Training; Post-infarction Nontraining: 39 postinfarction patients randomised to either a 3-month training group (n=20) or a nontraining group (n=19), and 19 normal controls.
- Healthy Controls: 19 age- and sex-matched healthy volunteers
Arm/Group | Post-infarction Training | Post-infarction Nontraining | Healthy Controls
Number analyzed (Participants) | 20 | 19 | 19
pg/ml
  Change of stromal-derived factor-1 | -196 (209) | -68 (175) | -57 (200)
  Change of vascular endothelial growth factor | 0.70 (1.41) | 0.95 (1.46) | -1.2 (2.92)
  Change of stem cell factor | 20 (120) | 17 (47) | -18 (60)

ADVERSE EVENTS:
Time Frame: Mean time from the onset of MI to initial evaluation was 8.3 (3.4) months. The groups did not differ in medication taken.No patients died, were hospitalized for coronary intervention, or had worsening symptoms during the 3-month study period.
Description: At baseline and the 3-month follow-up, all patients underwent a functional evaluation that included clinical evaluation, exercise testing, cardiac MRI and measurements of plasma angiogenic cytokines levels. Both groups were receiving stable and optimal pharmacological treatment supervised by their physicians.
Arm/Group | Postinfarction Training Patients | Postinfarction Nontraining Patients | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
First, our trial is small size. Second, these results are applicable only for male patients less than 65 years old with ST-segment elevation MI after successful PCI. Third, the source of angiogenic cytokines cannot be elucidated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No